CLINICAL TRIAL: NCT03644862
Title: A Prospective, Single Center, Non-comparative, 90-day Follow-up, Postmarket Clinical Investigation of Etafill in Patients With Cataract Surgery Via the Anterior Chamber
Brief Title: Study of Etafill in Patients With Cataract Surgery Via the Anterior Chamber
Status: Completed | Type: Observational
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CPH-401-201285
Record Dates: First submitted 2018-08-09; First posted 2018-08-23 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: etafill — Etafill is a HA formulation intended to be used in opthalmic anterior segment cataract surgery.

SUMMARY:
This prospective, single center, non-comparative, 90-day follow-up, post-market clinical investigation of etafill in patients undergoing cataract surgery.

The performance is measured by the preservation of endothelial cells measured by specular microscopy at the follow-up visit in comparison to baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for cataract surgery via the anterior chamber
* A negative urine pregnancy test at Visit 1 or 2
* Capability to understand information about the investigation, including patients' obligations, and willingness to take part, as evidenced by signed and dated informed consent

Exclusion Criteria:

* Patients with a known hypersensitivity to HA or other components of the device.
* Patients with corneal scars or corneal dystrophies interfering with study measurements
* Abnormal intraocular pressure which would interfere with surgery and follow up (in opinion of the investigator)
* Any other condition that in the opinion of the investigator would interfere with the participation in this investigation
* Any person dependent on the investigator or employees of the investigation site institution or the Sponsor.
* Current or previous (within 30 days of enrollment) treatment with another investigational drug and/or medical device or participation in another clinical study
* Patients whose participation in clinical trials is prohibited by the Austrian Medical Devices Act

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study patients will be recruited by the investigator, among patients scheduled to receive a standard cataract surgery taking inclusion and exclusion criteria into account. The investigator may also offer participation in the study to potential candidates identified in their patient database.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Specular microscopy to measure the preservation of endothelium cells | 90 days post surgery compared to baseline

SECONDARY OUTCOMES:
Specular microscopy to measure the corneal thickness | post surgery, 1 day and 90 days post surgery compared to baseline
Intraocular pressure measurement | post surgery, 1 day and 90 days post surgery compared to baseline
Questionnaire to assess the satisfaction with the application | day 0
  Questionnaire contains the subjective evaluation by the investigator of the IMD's rheological properties as well as the maintenance of the patient's anterior chamber and dome.
  Scale for the chamber and dome maintenance ranges from flat ( worst case) to full chamber (best case) maintained.
  Scale for rheological properties ranges from dispersive (worst case) to cohesive (best case).

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No